CLINICAL TRIAL: NCT00963313
Title: A 24 Week Open Label Study of the Utility of Adalimumab in Active Axial Forms of Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Dr. FRANCISCO J. BLANCO-GARCIA (Other)
Responsible Party: Sponsor-Investigator, Dr. FRANCISCO J. BLANCO-GARCIA, MD, PhD, Instituto de Investigacion Biomedica de A Coruna
Organization: Instituto de Investigacion Biomedica de A Coruna (Other)
Other Study IDs: SUE-ADA-2009-01
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Psoriatic Arthritis
Keywords: Axial psoriatic arthritis; Adalimumab; Humira; anti-TNF
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples recollected for analysing IL6 and MMP3 from patients blood serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab, injection: Adalimumab, one injection every fourteen days during 24 weeks.
  Interventions: Drug: Adalimumab (HUMIRA®)

INTERVENTIONS:
Drug: Adalimumab (HUMIRA®) — Prefilled syringes containing 40 mg Adalimumab in 0.8 ml injection solution. Study drug will be subcutaneously self-administered every 2 weeks during 24 weeks.
  Other Names: HUMIRA®

SUMMARY:
Based on published data and according to the approved product label for ankylosing spondylitis and psoriatic arthritis, it can be expected that adalimumab 40 mg every 14 days should be effective in psoriatic arthritic patients with axial involvement.

DETAILED DESCRIPTION:
A recent review from GRAPPA group evaluates therapies for PsA including peripheral and axPsA. Analysing particularly the results with present biologic therapies it has been proven that outcome data at 24 weeks show excellent results in the treatment of peripheral forms of PsA with either of the three biologics disposable in the market, that is to say infliximab, etanercept and adalimumab.

However when it comes to analyse data on PsA patients with axPsA there are not results at all. The design of clinical trials did not evaluate axial outcomes and therefore there is not a possibility of knowing whether these therapies are useful in axPsA.

This is an open label multicenter study designed to evaluate the effectivity of adalimumab 40 mg every 2 weeks during 24 weeks in patients with active axial PsA despite receiving Methotrexate, Sulfasalazine, Leflunomide or Cyclosporine, plus NSAIDs and no more than 10 mg of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 70 years.
* A negative pregnancy test for women of childbearing potential during the screening period.
* Subject must be evaluated for active or latent TB (tuberculosis) infection by using a PPD skin test (Mantoux test), Booster test, chest x-ray and detailed review of subjetc´s medical history.
* Subjects to whom the doctor has decided to prescribe adalimumab, because of fulfilling the requirements for this treatment.
* Diagnosed with PsA according to CASPAR criteria.
* Axial disease according to radiological criteria (at least unilateral sacroilitis grade II) and spinal inflammatory symptoms.
* Disease duration of no less than 24 weeks
* Patients with peripheral involvement (mixed forms of APs) must have been taking MTX for at least 12 weeks before screening and at stable doses of 10 to 25 mg/week for 8 weeks before screening, or salazopyrine up to 3 mg/daily, or cyclosporin 2mg/kg or leflunomide 20 mg daily in the same conditions as MTX.
* Patient's doses of NSAIDs and oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) should have been kept stable for 4 weeks before screening.

Exclusion Criteria:

* Contraindications for treatment with anti-TNF.
* Prior treatment with other TNF inhibitors or other investigational drugs during the last 30 days (etanercept 4 weeks, infliximab 8 weeks).
* Uncontrolled diabetes.
* Uncontrolled high blood pressure.
* Unstable ischemic heart disease.
* Congestive heart failure.
* Severe pulmonary disease.
* Chronic leg ulcer.
* History of cancer or malignant lymphoproliferative disease.
* Positive serology for Hepatitis B indicating active infection or positive serology for Hepatitis C.
* History of positive HIV status.
* Persistent, recurrent or severe infections requiring hospitalization or treatment with oral antibiotics within 14 days prior to enrollment.
* Previous diagnosis or signs highly indicative of central nervous system demyelinating diseases.
* Active tuberculosis, histoplasmosis or listeriosis.
* History or presence of confirmed blood dyscrasia.
* Female subjects who are pregnant or breast-feeding.
* History of clinically significant drug or alcohol abuse in the last year.
* Treatment with MTX, salazopyrine, ciclosporin or leflunomide initiated within the last 4 weeks before the screening. Treatment with corticosteroids (>10mg/day or equivalent or modified dose within the previous 4 weeks before screening). And patients where an intraarticular corticoid infiltration has been practised within the last 4 weeks before the screening will be excluded from the study.
* Treatment with more than one NSAID within the last 4 weeks before the screening.
* Patients treated with any DMARD different from MTX, cyclosporine, leflunomide and sulfasalazine.
* Dosage of concomitant MTX, cyclosporine, leflunomide and sulfasalazine must be stable during the study, otherwise it should be properly justified and recorded in the case report form.
* Patients treated with any analgesic different from acetominophen, NSAIDs, oxycodone, codeine, propoxyphene, tramadol, hydrocodone or combinations of these products or equivalents. The use of potent opioids is not permitted.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active axial forms of psoriatic arthritis
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
BASDAI score (Bath Ankylosing Spondylitis Disease Activity Index). | 12 WEEKS
  Proportion of patients that reach a BASDAI 50% at week 12, BASDAI 50% means an improvement from baseline of 50% or an improvement of two units on a 10 unit scale.
Number of participants with new adverse events. | 24 WEEKS

SECONDARY OUTCOMES:
ASAS 40 score. | 24 WEEKS
ASAS 50 and ASAS 70 score, 5/6. | 12 WEEKS
Evaluation of enthesitis. | 24 WEEKS
Peripheral articulation measured with DAS 28. | 24 WEEKS
Evaluation of extraarticular manifestations. | 24 WEEKS
Measure of laboratory parameters. | 24 WEEKS
  Hematology, biochemistry, CRP, ESR, HLA-B27 and rheumatoid factor.
Evaluation of quality of life. | 24 WEEKS
  SF36
Measure of PASI (Psoriasis Area and Severity Index). | 24 WEEKS
Measure of Modified NAPSI (Modified Nail Psoriasis Severity Index). | 24 WEEKS
Measure of BASFI (Bath Ankylosing Spondylitis Functioning Index). | 24 WEEKS
Evaluation of health. | 24 WEEKS
  HAQ (Health Assessment Questionarie).
Evaluation of dactylitis. | 24 WEEKS
Measure of inflammatory biomarkers (IL6 and MMP3). | 24 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Blanco-Garcia, MD, PhD, Study Chair — Complejo Hospitalario Universitario A Coruna
Locations (22):
- Spain (22):
  - Complejo Hospitalario Universitario A Coruna, A Coruña, A Coruna
  - Hospital Arquitecto Marcide-Novoa Santos, Ferrol, A Coruna
  - Hospital de Elche, Elche, Alicante
  - Hospital Comarcal Villajoyosa, Villajoyosa, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall d´Hebron, Barcelona, Barcelona
  - Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital Basurto, Bilbao, Bilbao
  - Hospital San Pedro de Alcantara, Cáceres, Caceres
  - Hospital General de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital Doctor Negrin, Las Palmas, Gran Canaria
  - Hospital Insular de Las Palmas, Las Palmas, Gran Canaria
  - Hospital Orense, Ourense, Orense
  - Hospital Pontevedra, Pontevedra, Pontevedra
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Monte Naranco, Oviedo, Principality of Asturias
  - Hospital de Salamanca, Salamanca, Salamanca
  - Hospital Donostia, Donostia / San Sebastian, San Sebastian
  - Hospital Virgen de la Macarena, Seville, Sevilla